CLINICAL TRIAL: NCT06880835
Title: INHALE-AIDEx: A Randomized Crossover Trial Evaluating the Effect of Inhaled Technosphere Insulin (Afrezza®) vs Rapid Acting Analogue Insulin on Exercise-Induced Hypoglycemia in Adults With Type 1 Diabetes Using Automated Insulin Delivery
Brief Title: Effect of Inhaled Technosphere Insulin vs RAA Insulin on Exercise-Induced Hypoglycemia in Adults With T1D Using Automated Insulin Delivery
Acronym: INHALE-AIDEx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Mannkind Corporation (Industry); Tandem Diabetes Care, Inc. (Industry); The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INHALE-AIDEx
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Exercise; Technosphere Insulin; Automated Insulin Delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Control IQ + sleep activity with TI (Experimental): TI for meal bolus with Control IQ + sleep activity pump setting
  Interventions: Device: Control IQ + sleep activity with TI
- Control IQ + sleep activity with Rapid-Acting Analogue (RAA) Comparator (No Intervention): RAA for meal bolus with with Control IQ + sleep activity pump setting
- Control IQ + exercise activity with Rapid-acting analogue (RAA) Control (No Intervention): RAA for meal bolus with Control IQ pump setting with transition to Control IQ + exercise activity pump setting one hour before start of exercise

INTERVENTIONS:
Device: Control IQ + sleep activity with TI — TI for meal bolus with Control IQ + sleep activity pump setting
  Arms: Control IQ + sleep activity with TI

SUMMARY:
This investigator-initiated study will enroll about 30 adults 18 to 65 years of age with type 1 diabetes (T1D) who are using the Tandem t:slim X2 insulin pump or Tandem Mobi insulin pump with Control-IQ or Control-IQ+ technology ("Control-IQ" which will refer to either Control-IQ or Control-IQ+). The study is being done to find out if inhaled insulin given for a meal is safer and better to use than a bolus of insulin through your pump when you exercise following a meal. Participants are asked to complete three study exercise visits in the clinic.

DETAILED DESCRIPTION:
The study is a 3-period randomized crossover trial, each with a structured afternoon exercise session following a standard lunch meal. The 3 sessions are as follows: (1) TI for meal bolus with pump in sleep mode, (2) RAA for meal bolus with pump in sleep mode, and (3) RAA for meal bolus with pump in standard mode with transition to exercise mode one hour before start of exercise. The study is being done to compare the efficacy and safety of TI versus RAA given as bolus for meal prior to initiating aerobic exercise in adults ≥18 to ≤ 65 years of age with T1D using Control-IQ.

All participants will complete 3 exercise sessions, with the order determined through randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent for study participation
2. Age ≥18 years to 65 years
3. Clinical diagnosis of T1D (per the Investigator)
4. Using Tandem t:slim X2 or Tandem Mobi insulin pump with Control-IQ for at least 90 days prior to screening visit
5. Using insulin aspart or insulin lispro in Tandem insulin pump
6. Total daily insulin dose 20 to 80 units
7. Usual RAA insulin bolus for 50 gram carbohydrate lunch meal is ≤12 units
8. Physically active, with at least 3 moderate or vigorous exercise sessions ≥30 minutes per typical week self-reported by participant
9. No medical, psychiatric, or other conditions, or medications being taken that in the Investigator's judgement would be a safety concern for participation in the study
10. No electrocardiogram (ECG) abnormality that in the judgment of the investigator, which will take into consideration the usual exercise performed by the participant and their overall medical condition, increases the risk of exercise
11. Investigator believes that the participant can safely follow the protocol
12. Able to read and understand written and spoken English or Spanish

Exclusion Criteria:

1. Use of inhaled insulin within one week prior to screening visit
2. History of asthma, chronic obstructive pulmonary disease (COPD), or any other clinically important pulmonary disease (e.g., cystic fibrosis or bronchopulmonary dysplasia), or significant congenital or acquired cardiopulmonary disease as judged by the Investigator
3. Smoking (includes cigarettes, cigars, pipes, marijuana, and vaping devices) within 90 days prior to screening visit and no plans to smoke during the study
4. History or current diagnosis of lung cancer
5. Forced expiratory volume in 1 second (FEV1) measurement of <70% of predicted Global Lung Function Initiative value
6. Pregnant or lactating, planning to become pregnant during the study, or is of childbearing potential and not on acceptable form of birth control (acceptable includes abstinence, condoms, oral/injectable contraceptives, IUD, or implant); childbearing potential means that menstruation has started, and the participant is not surgically sterile or greater than 12 months post-menopausal)

   • A pregnancy test is required for any person of childbearing potential.
7. An event of severe hypoglycemia, as judged by the Investigator, within the 90 days prior to screening visit
8. An episode of diabetic ketoacidosis (DKA) as defined in section 5.2 within the 90 days prior to screening visit
9. Any disease other than diabetes or current use (or anticipated use during the study) of any medication (e.g., beta blocker) that, in the judgment of the Investigator, may substantially impact glucose metabolism
10. Use of a non-insulin glucose-lowering medication (or weight-reduction medication with glucose-lowering effect) within 4 weeks prior to screening visit
11. Exposure to any investigational drug in the 90 days prior to the screening visit
12. Current or anticipated acute uses of oral, inhaled, or injectable glucocorticoids during the time period of the study (topical or intranasal glucocorticoid use is acceptable)
13. Current use of Hydroxyurea medication
14. Current or anticipated use of a low carbohydrate diet (<50 grams/day) or low calorie diet (<800 kcal/day) during the time period of the study
15. Current treatment for diabetic retinopathy
16. Known stage 4/5 chronic kidney disease or on dialysis
17. Having a direct supervisor at place of employment who is directly involved in conducting the clinical trial (as a study Investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Blood glucose <70 mg/dL | 90 minutes
  Blood glucose <70 mg/dL within 90 minutes from the start of exercise

OTHER OUTCOMES:
Exploratory Efficacy Outcome: Change in blood glucose from exercise start to nadir glucose | 90 minutes
  Change in blood glucose from exercise start to nadir glucose within 90 minutes from start of exercise
Exploratory Efficacy Outcome: Change in CGM glucose from exercise start to nadir glucose | 90 minutes
  Change in CGM glucose from exercise start to nadir glucose within 90 minutes from start of exercise
Exploratory Efficacy Outcome: Time in range 70-180 mg/dL | 90 minutes
  Time in range 70-180 mg/dL within 90 minutes from start of exercise
Exploratory Efficacy Outcome: Time in tight range 70-140 mg/dL | 90 minutes
  Time in tight range 70-140 mg/dL within 90 minutes from start of exercise
Exploratory Efficacy Outcome: Mean glucose | 90 minutes
  Mean glucose within 90 minutes from start of exercise
Exploratory Efficacy Outcome: CGM glucose <54 mg/dL | 90 minutes
  CGM glucose <54 mg/dL within 90 minutes from start of exercise
Exploratory Efficacy Outcome: CGM glucose <70 mg/dL | 90 minutes
  CGM glucose <70 mg/dL within 90 minutes from start of exercise
Exploratory Efficacy Outcome: CGM glucose >250 mg/dL | 90 minutes
  CGM glucose >250 mg/dL within 90 minutes from start of exercise
Exploratory Efficacy Outcome: CGM glucose >300 mg/dL | 90 minutes
  CGM glucose >300 mg/dL within 90 minutes from start of exercise
Safety Outcome: Severe hypoglycemia events | From enrollment to last clinic visit (up to ~12 weeks)
  Defined as events requiring assistance of another person due to cognitive impairment to actively administer carbohydrate, glucagon, or other resuscitative actions
Safety Outcome: Blood glucose <54 mg/dL during clinic | 210 minutes
  Blood glucose <54 mg/dL between start of meal and discharge from clinic
Safety Outcome: Blood glucose <70 mg/dL during clinic | 210 minutes
  Blood glucose <70 mg/dL between start of meal and discharge from clinic
Safety Outcome: Adverse events related to exercise procedure | From enrollment to last clinic visit (up to ~12 weeks)
  Adverse events related to the exercise procedure
Safety Outcome: Adverse events associated with technosphere insulin inhalation | From enrollment to last clinic visit (up to ~12 weeks)
  Adverse events associated with technosphere insulin (TI) inhalation: hypersensitivity reaction, acute bronchospasm, treatment provided for asthma symptoms, or other symptoms associated with TI dosing

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Rickels, MD, MA, Principal Investigator — University of Pennsylvania; Michael Ridell, PhD, Study Chair — York University
Locations (3):
- United States (3):
  - University of Louisville, Louisville, Kentucky
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided
A limited dataset is expected to be made available.